CLINICAL TRIAL: NCT01447524
Title: Very Low Calorie Diet: a Quick Therapeutic Tool to Improve Beta Cell Function in Morbidly Obese Patients With Type 2 Diabetes Mellitus
Brief Title: Caloric Restriction and Insulin Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Simona Frontoni, MD, PhD, University of Rome Tor Vergata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48/2009
Record Dates: First submitted 2011-09-30; First posted 2011-10-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Morbid Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Very Low Calorie Diet — Very Low Calorie Diet consisted of a 400 kcal/day diet, with percentage distribution of lipids, proteins and carbohydrates, according to Italian Standards of Care.

SUMMARY:
Caloric restriction in obese diabetic patients quickly improves glucose control, independently from weight loss. However, the early effects of a very-low calorie diet (VLCD) on insulin sensitivity and insulin secretion in morbidly obese patients with type 2 diabetes are still unclear.

The objective of this study was to investigate the relative contributions of insulin sensitivity and/or secretion to the improvement in glucose metabolism, after one week of caloric restriction, in severely obese diabetic patients.

For this purpose, hyperglycemic clamps were performed in 14 severely obese (BMI> 40 kg/m2) patients with type 2 diabetes in good glucose control (HbA1c <7.5%), before and after 7 days on VLCD 400 kcal/day.

DETAILED DESCRIPTION:
In obese patients with type 2 diabetes mellitus, lifestyle modifications resulting in weight loss improve or even normalize blood glucose. This beneficial effect on glucose control is accounted for by improvements in both insulin secretion and insulin sensitivity. However, the metabolic effects of caloric restriction per se may be, at least in part, independent of body weight reduction. Furthermore, improved control of blood glucose in type 2 diabetes by very low calorie diet (VLCD) for 40 days was documented during the first 10 days of caloric restriction, when weight loss was still trivial. When caloric intake was increased after weight reduction, plasma glucose increased in spite of no weight rebound. The mechanism(s) underlying these early improvements caused by a VLCD in patients with type 2 diabetes have been assessed only in a few studies. Thus, a fall in hepatic glucose production and a modest increase in insulin sensitivity were reported as early as 7 days after a very low calorie diet. A subsequent study replicated the effects of short term VLCD on hepatic glucose production, but not on whole body insulin sensitivity.

As to beta cell function, earlier studies reported an apparent improvement in insulin secretion rate during the oral glucose tolerance test (OGTT), after short-term application of a VLCD. However, no formal investigation of beta cell sensitivity to glucose was performed, and, since glucose was given per os, other factors (e.g. incretins, ghrelin) might have been involved. One study reported an improvement of beta cell response during hyperglycemic clamps, i.e. excluding gut related factors, after 8 weeks of a VLCD and during a weight stabilization period, i.e. in the absence of the negative energy balance signal. Furthermore, by study design, it did not explore the first phase secretory response to glucose.

Quite recently, Lim and coll. reported that, in patients with type 2 diabetes, a VLCD markedly improved glucose control in a few days, and that ameliorations of both liver insulin sensitivity and beta cell sensitivity to glucose were the mechanisms primarily involved. Prolongation of the VLCD for 8 weeks led to an apparent remission of diabetes. This and most of earlier mechanistic studies were performed in patients with BMI around 30-35, in whom, according to most current guidelines, metabolic surgery should not be considered a treatment option. In patients with type 2 diabetes undergoing bariatric surgery, improvements in glucose control and in beta cell function are detectable before a significant weight loss occurred, and there is a strong suggestion that intestinal bypass procedures may have metabolic effects (e.g. on beta cell) that are independent of their effect on body weight, possibly involving the incretin axis. Furthermore, remission rates of type 2 diabetes following bariatric surgery as high as 70-80% have been reported.

Thus, it would be important to know whether in severely obese patients with type 2 diabetes, who are potential candidates for metabolic surgery, a short term VLCD exerts effects similar to those reported in less obese patients.

The investigators therefore performed a preliminary proof-of-concept study to assess whether in severely obese patients with type 2 diabetes 7 days of VLCD affect glucose control through changes in either beta cell function or insulin sensitivity or both.

Participants were studied at baseline and then after 7 days of caloric restriction (VLCD). VLCD consisted of a 400 kcal/day diet, with percentage distribution of lipids, proteins and carbohydrates, according to Italian Standards of Care.

Both at baseline and at the end of VLCD, a hyperglycemic insulin clamp study was performed in all patients, as previously described. All studies were carried out at 08.00, after a 12-hour overnight fast, while the subjects were lying in bed, and lasted 180'. In all subjects two intravenous catheters were inserted into an ante-cubital vein and (retrogradely) into a wrist vein for substance infusion and sampling of arterialized blood, respectively, according to the hot box technique. After a 60 min period to establish baseline (-60'- 0'), at time 0' a hyperglycemic glucose clamp was carried out for the following 120', as previously described. Plasma glucose was measured at bedside every 2'-5' as needed and was clamped at 7.0 mmol/L (126 mg/dl) above baseline values. Under these conditions of constant hyperglycemia, the normal beta cell secretory response is biphasic with an early burst of insulin release within the first 10 minutes (first phase), followed by a later monotonically increasing hormone release (second phase).

Blood samples for glucose, C-peptide and insulin determinations were drawn every 2.5 min from 0 to 15 min and every 15 min from 15 to 120 min.

The acute insulin response (AIR) was calculated as the average incremental plasma insulin concentration at 2.5, 5.0, 7.5 and 10 min of the hyperglycemic clamp.

Second phase insulin response (2ndIR) was computed as the average incremental insulin concentration between 60' and 120' of the hyperglycemic clamp.

Glucose disposal during the clamp was computed as the rate of exogenous glucose infusion corrected for the (minimal) changes in the glucose pool (M value; units: µmol.min-1.m-2 BSA).

The metabolic clearance rate of glucose during the clamp was computed as the ratio between the M value and the prevalent glucose concentration. Under these experimental conditions, the metabolic clearance rate of glucose is a direct experimental measurement of the Disposition Index of second phase insulin secretion (DI; units: ml. min-1.m-2 BSA), in that it is the whole body use of glucose achieved by the beta cell at the same experimentally fixed glucose concentration. It measures whole body capability to dispose an intravenous glucose load, and it reflects beta cell adequacy to adjust to prevailing insulin resistance and insulin clearance. This DI has two advantages: 1. It is a direct experimental measure, not the product of two different experimental assessments; 2. At variance with all other DIs, it requires no assumptions regarding the mathematical relationship linking insulin sensitivity to beta cell secretory response or glucose-stimulated insulin concentrations.

Insulin sensitivity during the hyperglycemic clamp was calculated as the ratio of metabolic clearance rate of glucose divided by the average insulin concentration achieved between 60' and 120' (IS; units: [(ml. min-1.m-2 BSA)/ (pmol/L)].

The analyses of the glucose and C-peptide curves during the hyperglycemic clamp follow the general strategy proposed by several laboratories with some slight modifications, which have been previously described in detail.

The main outputs of this model are:

1. First phase parameters

   * Total amount of insulin secreted due to first phase (1stISR; units: pmol.m-2 BSA)
   * Glucose sensitivity of first phase secretion (σ1), expressed as the amount of insulin secreted in response to a rate of increase in glucose concentration of 1 mmol/liter between time 0 and 1 min of the study (units: [(pmol.m-2 BSA)/(mM.min-1)]
2. Second phase parameters

   * Total amount of insulin secreted due to second phase (2ndISR; units: pmol.m-2 BSA);
   * Glucose sensitivity of second-phase secretion (σ2), expressed as the steady-state insulin secretion rate in response to a step increase in glucose concentration of 1 mmol/liter above baseline (units: [(pmol.min-1.m-2 BSA/(mmol/L)].

Finally, an index of insulin clearance (InsClearIndex; units: L.min-1.m-2 BSA) was calculated as the ratio of the average insulin secretion rate divided by the average insulin concentration during the hyperglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* diet or oral hypoglycaemic agents
* morbid obesity (BMI > 40kg/m2)
* good metabolic control (HbA1C <7.5%)

Exclusion Criteria:

* treatment with GLP-1 agonists, DPP-4 inhibitors, insulin
* serum creatinine >150 µmol/l

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin sensitivity at 7 days | At baseline and after 7 days of Very Low Calorie Diet
  Insulin sensitivity was measured at baseline (hospital entry) and after a 7 day very low calorie diet.
Change from baseline in insulin secretion at 7 days. | At baseline and after 7 days of Very Low Calorie Diet
  Insulin secretion was measured at baseline (hospital entry) and after a 7 day very low calorie diet.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Frontoni, MD, PhD, Study Chair — University of Rome Tor Vergata- Diabetes, Fatebenefratelli Hospital, Rome
Locations (1):
- San Giovanni Calibita Fatebenefratelli Hospital, Rome, Italy

REFERENCES:
- [Background] UK Prospective Diabetes Study 7: response of fasting plasma glucose to diet therapy in newly presenting type II diabetic patients, UKPDS Group. Metabolism. 1990 Sep;39(9):905-12. PMID 2392060
- [Background] Henry RR, Scheaffer L, Olefsky JM. Glycemic effects of intensive caloric restriction and isocaloric refeeding in noninsulin-dependent diabetes mellitus. J Clin Endocrinol Metab. 1985 Nov;61(5):917-25. doi: 10.1210/jcem-61-5-917. PMID 4044780
- [Background] Taylor R. Pathogenesis of type 2 diabetes: tracing the reverse route from cure to cause. Diabetologia. 2008 Oct;51(10):1781-9. doi: 10.1007/s00125-008-1116-7. Epub 2008 Aug 26. PMID 18726585
- [Background] Wing RR, Blair EH, Bononi P, Marcus MD, Watanabe R, Bergman RN. Caloric restriction per se is a significant factor in improvements in glycemic control and insulin sensitivity during weight loss in obese NIDDM patients. Diabetes Care. 1994 Jan;17(1):30-6. doi: 10.2337/diacare.17.1.30. PMID 8112186
- [Background] Kelley DE, Wing R, Buonocore C, Sturis J, Polonsky K, Fitzsimmons M. Relative effects of calorie restriction and weight loss in noninsulin-dependent diabetes mellitus. J Clin Endocrinol Metab. 1993 Nov;77(5):1287-93. doi: 10.1210/jcem.77.5.8077323.
- [Background] Lara-Castro C, Newcomer BR, Rowell J, Wallace P, Shaughnessy SM, Munoz AJ, Shiflett AM, Rigsby DY, Lawrence JC, Bohning DE, Buchthal S, Garvey WT. Effects of short-term very low-calorie diet on intramyocellular lipid and insulin sensitivity in nondiabetic and type 2 diabetic subjects. Metabolism. 2008 Jan;57(1):1-8. doi: 10.1016/j.metabol.2007.05.008. PMID 18078853
- [Background] Markovic TP, Jenkins AB, Campbell LV, Furler SM, Kraegen EW, Chisholm DJ. The determinants of glycemic responses to diet restriction and weight loss in obesity and NIDDM. Diabetes Care. 1998 May;21(5):687-94. doi: 10.2337/diacare.21.5.687. PMID 9589225
- [Background] Gumbiner B, Polonsky KS, Beltz WF, Griver K, Wallace P, Brechtel G, Henry RR. Effects of weight loss and reduced hyperglycemia on the kinetics of insulin secretion in obese non-insulin dependent diabetes mellitus. J Clin Endocrinol Metab. 1990 Jun;70(6):1594-602. doi: 10.1210/jcem-70-6-1594. PMID 2189885
- [Background] Lim EL, Hollingsworth KG, Aribisala BS, Chen MJ, Mathers JC, Taylor R. Reversal of type 2 diabetes: normalisation of beta cell function in association with decreased pancreas and liver triacylglycerol. Diabetologia. 2011 Oct;54(10):2506-14. doi: 10.1007/s00125-011-2204-7. Epub 2011 Jun 9. PMID 21656330
- [Background] American Diabetes Association. Standards of medical care in diabetes--2011. Diabetes Care. 2011 Jan;34 Suppl 1(Suppl 1):S11-61. doi: 10.2337/dc11-S011. No abstract available. PMID 21193625
- [Background] Mingrone G, Castagneto-Gissey L. Mechanisms of early improvement/resolution of type 2 diabetes after bariatric surgery. Diabetes Metab. 2009 Dec;35(6 Pt 2):518-23. doi: 10.1016/S1262-3636(09)73459-7. PMID 20152737
- [Background] Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. Am J Med. 2009 Mar;122(3):248-256.e5. doi: 10.1016/j.amjmed.2008.09.041. PMID 19272486
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2010 Jan;33 Suppl 1(Suppl 1):S62-9. doi: 10.2337/dc10-S062. No abstract available. PMID 20042775
- [Background] Bruno G, De Micheli A, Frontoni S, Monge L; Societa Italiana di Diabetologia-Associazione Medici Diabetologi (SID-AMD) Working Group on the Standards of Care for Diabetes. Highlights from "Italian Standards of care for Diabetes Mellitus 2009-2010". Nutr Metab Cardiovasc Dis. 2011 Apr;21(4):302-14. doi: 10.1016/j.numecd.2010.08.009. Epub 2010 Sep 18. PMID 20851582
- [Background] Allain CC, Poon LS, Chan CS, Richmond W, Fu PC. Enzymatic determination of total serum cholesterol. Clin Chem. 1974 Apr;20(4):470-5. No abstract available. PMID 4818200
- [Background] Bucolo G, David H. Quantitative determination of serum triglycerides by the use of enzymes. Clin Chem. 1973 May;19(5):476-82. No abstract available. PMID 4703655
- [Background] Weykamp C, John WG, Mosca A. A review of the challenge in measuring hemoglobin A1c. J Diabetes Sci Technol. 2009 May 1;3(3):439-45. doi: 10.1177/193229680900300306. PMID 20144280
- [Background] Racette SB, Weiss EP, Villareal DT, Arif H, Steger-May K, Schechtman KB, Fontana L, Klein S, Holloszy JO; Washington University School of Medicine CALERIE Group. One year of caloric restriction in humans: feasibility and effects on body composition and abdominal adipose tissue. J Gerontol A Biol Sci Med Sci. 2006 Sep;61(9):943-50. doi: 10.1093/gerona/61.9.943. PMID 16960025
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] SCHMIDT FH. [Enzymatic determination of glucose and fructose simultaneously]. Klin Wochenschr. 1961 Dec 1;39:1244-7. doi: 10.1007/BF01506150. No abstract available. German. PMID 14498709
- [Background] Pfutzner A, Lobig M, Fortunato A, Forst T. Evaluation of a new fully automated one-step C-peptide chemiluminescence assay (LIAISON C-Peptid). Clin Lab. 2003;49(5-6):227-32. PMID 15285178
- [Background] Sapin R. Insulin assays: previously known and new analytical features. Clin Lab. 2003;49(3-4):113-21. PMID 12705692
- [Background] Mari A, Ahren B, Pacini G. Assessment of insulin secretion in relation to insulin resistance. Curr Opin Clin Nutr Metab Care. 2005 Sep;8(5):529-33. doi: 10.1097/01.mco.0000171130.23441.59. PMID 16079624
- [Background] Cobelli C, Toffolo GM, Dalla Man C, Campioni M, Denti P, Caumo A, Butler P, Rizza R. Assessment of beta-cell function in humans, simultaneously with insulin sensitivity and hepatic extraction, from intravenous and oral glucose tests. Am J Physiol Endocrinol Metab. 2007 Jul;293(1):E1-E15. doi: 10.1152/ajpendo.00421.2006. Epub 2007 Mar 6. PMID 17341552
- [Background] Cali' AM, Bonadonna RC, Trombetta M, Weiss R, Caprio S. Metabolic abnormalities underlying the different prediabetic phenotypes in obese adolescents. J Clin Endocrinol Metab. 2008 May;93(5):1767-73. doi: 10.1210/jc.2007-1722. Epub 2008 Feb 26. PMID 18303080
- [Derived] Malandrucco I, Pasqualetti P, Giordani I, Manfellotto D, De Marco F, Alegiani F, Sidoti AM, Picconi F, Di Flaviani A, Frajese G, Bonadonna RC, Frontoni S. Very-low-calorie diet: a quick therapeutic tool to improve beta cell function in morbidly obese patients with type 2 diabetes. Am J Clin Nutr. 2012 Mar;95(3):609-13. doi: 10.3945/ajcn.111.023697. Epub 2012 Feb 8. PMID 22318758